CLINICAL TRIAL: NCT06402929
Title: Self-stigma and Strategic Disclosure Amongst Canadian Postsecondary Students
Brief Title: Honest, Open, Proud - College for Post-Secondary Students With Mental Health Challenges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lakehead University (Other)
Collaborators: Illinois Institute of Technology, Chicago, USA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1468496
Record Dates: First submitted 2024-05-03; First posted 2024-05-07 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Stigmatization; Mental Health Issue; Disclosure
Keywords: Mental Illness; Stigma; Self-Stigma; Post-Secondary Students; Group Intervention; Disclosure
MeSH Terms: conditions — Stereotyping; Mental Disorders; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Honest Open Proud - College (HOP-C) (Experimental)
  Interventions: Behavioral: Honest Open Proud - College (HOP-C)
- Waitlist Control (No Intervention): Participants randomized to the waitlist control condition complete the study measures at the same timepoints as the experimental group while remaining on a waiting list for the program. Following this, participants randomized to the waitlist are invited to participate in HOP-C without completing study measures.

INTERVENTIONS:
Behavioral: Honest Open Proud - College (HOP-C) — The program consists of three weekly workshops that are two hours in duration. There is a fourth booster workshop (two hours in duration) one month following program completion. All workshops will be held over an online videoconferencing platform.
  HOP-C is a group program led by trained peer facilitators who have lived mental illness experience. Major topics that the program covers are:
  1. discussing different types of disclosure;
  2. conducting a cost-benefit analysis of disclosing in different situations;
  3. strategies to anticipate how certain people will respond to disclosure when deciding on who to disclose to;
  4. disclosure via social media; and
  5. a guided creation of participants' own disclosure narrative.
  During the booster workshop, participants will be encouraged to reflect on their disclosure decisions, and periodically revisit their disclosure cost-benefit analysis in deciding if and when to disclose in the future.
  Arms: Honest Open Proud - College (HOP-C)

SUMMARY:
The purpose of the study is to evaluate the efficacy of an online format of the group-based intervention "Honest Open Proud-College" among Canadian post-secondary students.

DETAILED DESCRIPTION:
Mental health issues have been highlighted as a growing concern within the post-secondary student population. Studies show that one significant concern for post-secondary students pertains to disclosing their mental challenges to others. Disclosure decisions are especially relevant for postsecondary students in the context of academic and social support. Students with mental health challenges who do not receive helpful accommodations may experience greater stress related to academics. Students also note that, in navigating their social sphere, they often need to consider what aspects of their mental health challenges to share in what situations.

As such, students often need to make decisions about whether to conceal or disclose their mental health challenges, both of which have their own pros and cons. Disclosure is a complex decision that requires consideration of personal and contextual factors. Honest, Open, Proud-College (HOP-C) is a peer-led, group-based intervention, that supports post-secondary students in the process of making decisions to disclose their mental health conditions. This study will evaluate the impacts of HOP-C administered through a videoconferencing platform on personal, social, and disclosure related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age 17 to 29 years old
* Enrolment in an university or college in Canada
* Self-identify as experiencing mental health challenges
* Moderate level of self-reported self-stigma (score 4 or higher on the screening item "Do you feel ashamed about dealing with anxiety, depression, or any other mental health challenges?", rated from 1, not at all, to 7, very much)

Exclusion Criteria:

-

Ages: 17 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Self-Stigma of Mental Illness Scale-Short Form (Corrigan et al., 2012) | Baseline, Post Intervention (3 weeks), and Post Booster (7 weeks)
Attitudes to Disclosure Questionnaire (Mayer et al., 2022) | Baseline, Post Intervention (3 weeks), and Post Booster (7 weeks)
Empowerment Scale (Rogers et al., 1997) | Baseline, Post Intervention (3 weeks), and Post Booster (7 weeks)

SECONDARY OUTCOMES:
Stigma Stress Scale (Rüsch, Corrigan, Powell, et al., 2009; Rüsch, Corrigan, Wassel, et al., 2009) | Baseline, Post Intervention (3 weeks), and Post Booster (7 weeks)
Rosenberg Self-Esteem Scale (Rosenberg, 1965) | Baseline, Post Intervention (3 weeks), and Post Booster (7 weeks)
Self-Efficacy about Disclosure Scale (Conley et al., 2019; Rüsch et al., 2014) | Baseline, Post Intervention (3 weeks), and Post Booster (7 weeks)
Multidimensional Scale of Perceived Social Support (Zimet et al., 1988) | Baseline, Post Intervention (3 weeks), and Post Booster (7 weeks)
General Help Seeking Questionnaire (Wilson et al., 2005) | Baseline, Post Intervention (3 weeks), and Post Booster (7 weeks)
Actual Help Seeking Questionnaire (Rickwood et al., 2005) | Baseline, Post Intervention (3 weeks), and Post Booster (7 weeks)

OTHER OUTCOMES:
Depression-Anxiety-Stress Scale-21 (DASS-21; Lovibond & Lovidbond, 1995) | Baseline, Post Intervention (3 weeks), and Post Booster (7 weeks)
Online Experience Questionnaire | Post Intervention (3 weeks)
  Assesses participants' experience with HOP-C in an online format. Consists of 10 items asking about comfortability and presentation of session content over the video conferencing platform. There is an additional question welcoming other comments and concerns.
Disclosure Worksheet | Post Intervention (3 weeks) and Post Booster (7 weeks)
  Assess disclosure behaviours using the "Details of Your Disclosure- How Did it Go?" Worksheet in the HOP-C manual. This worksheet collects information on whether the participant disclosed, who they disclosed to, and the participant's self-reported satisfaction with the exchange and the positivity of the exchange.

CONTACTS AND LOCATIONS:
Locations (1):
- Lakehead University, Thunder Bay, Ontario, Canada